CLINICAL TRIAL: NCT00462254
Title: Ramelteon (ROZEREM) in the Treatment of Sleep Disturbances Associated With Parkinson's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study discontinued.
Sponsor: Southern California Institute for Research and Education (Other)
Responsible Party: Andrius Baskys, M.D., VA Long Beach Healthcare System
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #789
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Parkinson's Disease
Keywords: Ramelteon; Parkinson's disease; Sleep disturbances
MeSH Terms: conditions — Parkinson Disease; Parasomnias | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Day 1-3: placebo run-in - 8 mg of placebo orally 30 minutes before bedtime. Days 4-11: true drug - 8 mg of Ramelteon orally 30 minutes before bedtime. Days 12-14: crossover - 8 mg of placebo orally 30 minutes before bedtime. Days 15-22: continue placebo.
  Interventions: Drug: ROZEREM
- B (Other): Day 1-3: Placebo run-in - 8 mg of placebo orally 30 minutes before bedtime. Days 4-11: continue placebo. Days 12-14: crossover - 8 mg of placebo orally 30 minutes before bedtime. Days 15-22: true drug - 8 mg of Ramelteon orally 30 minutes before bedtime.
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: ROZEREM — 8 mg tablet orally 30 minutes before bedtime for 8 days (Days 4-11).
  Other Names: Ramelteon
  Arms: A
Drug: Ramelteon — 8 mg tablet orally 30 minutes before bedtime for 8 days (Days 15-22).
  Other Names: Rozerem
  Arms: B

SUMMARY:
Patients with Parkinson's disease represent a significant proportion of VA elderly patients. Sleep disturbances and caregiver burnout association with this condition represent a significant problem. In this study, the investigators propose to perform an evaluation of a fixed doe of ramelteon on sleep in VA outpatients diagnosed with Parkinson's disease.

The hypothesis to be examined is that ramelteon will improve the quality of sleep in patients with Parkinson's disease while indirectly improving the quality of life for the patients and caregivers. The investigators further hypothesize that these changes will occur through restructuring and normalization of the sleep architecture.

DETAILED DESCRIPTION:
It is well established that sleep disturbances are common in patients with neurodegenerative disorders such as Parkinson's disease. Together with psychosis and other behavioral abnormalities they contribute to the stress, anxiety and cognitive decline of patients, caregiver burnout and depression, as well as health care provider frustration. The mechanisms of the sleep disturbances in these conditions are still poorly understood and no rational or effective treatments have been proposed. Recent data from a study of ramelteon in the elderly showed a striking ability of this compound to improve quality of sleep disturbances in Parkinson's disease.

Objectives of this study are:

* To examine the effects of ramelteon on the quality of sleep using sleep evaluation instruments (SDQ-Sleep Disorder Questionnaire and Neuropsychiatric Inventory with Caregiver Distress (NPI-D) Sleep Behavior Subscale administered to the patient and/or their bed partner.
* To examine the effects of ramelteon on daytime sleepiness and memory using Epworth Sleepiness Scale (ESS) and Hopkins Verbal Learning Test (HVLT).
* To examine the effects of ramelteon on the sleep/wake cycle and day/night activity patterns over a prolonged period of time (1 week) using a motion logger (continuous motor activity recording device) and computerized data analysis.
* To examine the effects of ramelteon on sleep architecture in a sample of patients with confirmed sleep disturbance, before and after ramelteon treatment by using polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* 45-85 years of age and living in the community
* Male or female of non-child bearing potentials (non-child bearing is defined as at lease 6 months post-menopause or surgically sterile)
* Must have a diagnosis of Parkinson's disease
* Must have complaints of sleep disturbance

Exclusion Criteria:

* Patients with diagnosis of or those meeting DSM-IV criteria for major depression, schizophrenia or schizoaffective disorder, bipolar disorder, substance abuse disorder, other mental illness that is known to contribute to sleep disturbance, epilepsy, other medical conditions that are known to cause or contribute to sleep disturbances
* Patients currently using melatonin or ramelteon, hypnotics, benzodiazepines, antidepressants, blood-brain barrier permeable beta blockers, steroids, antipsychotics
* Patients with clinically significant blood or urine abnormalities
* Patients who have taken any investigational drug less than 1 month prior to the baseline visit
* Patients with multiple concomitant disorders with or without medications thought to produce sleep disturbances
* Patients with pre-existing sleep disturbances unrelated to Parkinson's disease
* Patients with severe hepatic impairment (Child-Pugh Class C)
* Patients with severe COPD (those with elevated pCO2 levels or those needing nocturnal oxygen therapy
* Patients with severe sleep apnea
* Patients who have sensitivity to ramelteon or any constituents of the Rozerem preparation
* Patients taking rifampin or potent inducers of CYP1A2, CYP3A4, CYP2C9 (ketoconazole, fluconazole)
* Patients living in a nursing home. Those living in assisted living facilities and board and care facilities may be included
* Patients unable to comply with the study protocol

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory with Caregiver Distress (NPI-D) Sleep Behavior Subscale | One and one-half years
The Epworth Sleepiness Scale | One and one-half years
Sleep Disorders Questionnaire (short form) | One and one-half years

SECONDARY OUTCOMES:
Memory - Hopkins Verbal Learning Test (HVLT) | One and one-half years
Movement - Abnormal Involuntary Movement Scale (AIMS) | One and one-half years
Movement - Unified Parkinson's Disease Rating Scale (UPDRS) | One and one-half years
Movement - Continuous motor activity (actigraphy/motion logger) | One and one-half years

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Baskys, M.D., Principal Investigator — VA Long Beach Healthcare System
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- See also: Southern California Institute for Research and Education website — http://www.scire-lb.org